CLINICAL TRIAL: NCT00185185
Title: Multi-Centre Olmesartan Atherosclerosis Regression Evaluation (MORE)
Brief Title: Olmesartan Medoxomil in Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Responsible Party: Petra Laeis, Daichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-866/27
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Essential Hypertension; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Essential Hypertension; Atherosclerosis | interventions — Olmesartan Medoxomil; Atenolol; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): olmesartan medoxomil
  Interventions: Drug: Olmesartan medoxomil; Drug: Hydrochlorothiazide
- 2 (Active Comparator): atenolol
  Interventions: Drug: Atenolol; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil
  Arms: 1
Drug: Atenolol
  Arms: 2
Drug: Hydrochlorothiazide — tablets
Drug: olmesartan medoxomil — tablets
  Arms: 1
Drug: atenolol — tablets
  Arms: 2

SUMMARY:
This is a study in hypertensive patients with atherosclerosis and increased cardiovascular risk. The efficacy of olmesartan medoxomil on atherosclerosis is measured.

ELIGIBILITY:
Inclusion Criteria:

* Mean sitting sBP and dBP prior to randomization of 140-180/90-105 mmHg
* Increased cardiovascular risk, e.g.: a) documented or clinical signs of peripheral atherosclerotic disease stage IIa or lower; b) diabetes mellitus type 2; c) left ventricular hypertrophy on echo; d) current smoking; e) old myocardial infarction, stroke or TIA
* Intima-media thickness of the common carotid artery greater than or equal to 0.8 and less than or equal to 1.6 mm (measured ultrasonographically) or the plaque volume of the carotid bulb greater than or equal to 4 μl and less than or equal to 500 μl

Exclusion Criteria:

* Body mass index > 30
* Any type of known secondary hypertension
* Electrocardiographic evidence of 2nd or 3rd degree atrioventricular block, atrial fibrillation, cardiac arrhythmia requiring therapy or bradycardia at rest (< 50/min)
* Obstructive pulmonary disease
* Claudicatio intermittens
* History or clinical evidence of any significant gastrointestinal, respiratory, hematological, metabolic, immunological or any other underlying disease which in the opinion of the investigator would interfere with the patient's participation in the trial
* Hypersensitivity or contraindication to ARBs, Beta-Blockers, HCTZ or any cross allergy
* Pre-treatment with ARBs or ACE inhibitors within 6 months prior to screening
* Treatment with disallowed medication
* Pregnant or breastfeeding females or females of childbearing potential without adequate contraception
* History of alcohol and/or drug abuse

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2001-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change of intima media thickness of the common carotid artery on the leading side of the neck.

SECONDARY OUTCOMES:
-Change in plaque volume in the common carotid artery or the carotid bulb.
-Change of intima media thickness of the common carotid artery.
-Changes of diastolic and systolic blood pressure.
-Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Klaus O Stumpe, MD, Principal Investigator — Medizinische Poliklinik der Friedrich-Wilhelms-Universitat, Bonn, Germany
Locations (1):
- Munich, Germany

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307